CLINICAL TRIAL: NCT01817101
Title: Field Trial With Omega-3 Fatty Acid Supplementation for the Prevention of Cognitive Decline in a Very Elderly Population
Brief Title: Dietary Supplement for the Prevention of Cognitive Decline in a Very Elderly Population.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DIET
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2013-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Supplement capsule (Active Comparator): One capsule at meals (3 each day) during 1 year with Omega-3 fatty acid supplementation
  Interventions: Dietary Supplement: Omega-3 fatty acid supplementation
- Empty gelatine capsule (Placebo Comparator): One capsule at meals (3 each day during 1 year)

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid supplementation — Gelatine capsule, 1 at each meals (3 per day) during one year
  Arms: Dietary Supplement capsule

SUMMARY:
The purpose of this study is to determine whether an omega-3 fatty acid supplementation is effective in the prevention of progressive cognitive decline in elderly people aged 75 years or older.

DETAILED DESCRIPTION:
Participants are residents at three nursing homes in Pamplona (Spain). We assumed that 20% of elderly people have a cognitive decline and we estimated a 5% of cognitive decline in the intervention group. Sample size estimated was 85 participants for each arm, assuming two groups with an alpha of 0.05, 80% power and accounting for 10% of participants lost to follow-up.

Repeated measures ANOVA, Cox regression and multiple linear regression analysis will be used for the statistical analysis of data.

ELIGIBILITY:
Inclusion Criteria:

* Elderly people aged 75 years or older
* Global Deterioration Scale < 4
* Capacity to complete the tests

Exclusion Criteria:

* Neurological, physical or psychiatry conditions, obtained from the medical history, that may have an influence on the cognitive function.
* Dementia
* History of epilepsy, convulsions

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination | Six months / one year
  MMSE is a brief questionnaire test that is used to screen for cognitive impairment. A validated test in Spanish will be used:
  Lobo A. Saza P. Marcos G, Díaz J, De la Cámara C, Ventura T et al: Revalidación y normalización del Mini-Examen Cogniscitivo (primera versión en castellano del Mini-Mental Status Examination) en la población general geriátrica. Med Clin (Barc) 1999;112:767-774.

SECONDARY OUTCOMES:
Short Portable Mental Status Questionnaire (SPMSQ) | One year
  A questionnaire for the assessment of organic brain deficit in elderly patients (Pfeiffer E. A short portable mental status questionnaire for the assessment of organic brain deficit in elderly patients. J Am Geriatr Soc. 1975;23:433-41)
Verbal fluency test | One year
  Category verbal fluency test. Rosen W.: "Verbal fluency in aging and dementia". J. Clin Neuropsychol 1980;2: 135-146.
Clock-drawing test | One year
  A cognitive test that covers a wide range of cognitive function. Battersby, W.S., Bender, M.B., Pollack, M. y Kahn, R.L. Unilateral "spatial agnosia" ("inattention") in patients with cortical lesions. Brain 1956; 79: 68-93.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin Baleztena, MD, Principal Investigator — Clinica Universidad de Navarra
Locations (3):
- Spain (3):
  - Amma Argaray, Pamplona, Navarre
  - AMMA Mutilva, Pamplona, Navarre
  - AMMA Oblatas, Pamplona, Navarre